CLINICAL TRIAL: NCT02601313
Title: A Phase 2 Multicenter Study Evaluating the Efficacy of KTE-X19 in Subjects With Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Study of Brexucabtagene Autoleucel (KTE-X19) in Participants With Relapsed/Refractory Mantle Cell Lymphoma (Cohort 1 and Cohort 2)
Acronym: ZUMA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTE-C19-102; 2015-005008-27 (EudraCT Number); 2023-506641-35 (Other: European Medicines Agency)
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Relapsed/Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — brexucabtagene autoleucel; Cyclophosphamide; fludarabine; axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axicabtagene ciloleucel/brexucabtagene autoleucel (KTE-X19) (Experimental): Participants with relapsed/refractory mantle cell lymphoma (MCL) will receive conditioning chemotherapy (CTE) consisting of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day intravenous (IV) infusion for 3 days followed by a single infusion of axicabtagene ciloleucel at a targeted dose of 2 x 10^6 anti-CD19 chimeric antigen receptor (CAR) T cells/kg on Day 0 or brexucabtagene autoleucel (KTE-X19) at a targeted dose of 2 x 10^6 CAR T cells/kg, with a maximum dose of 2 x 10^8 anti-CD19 CAR T cells for participants ≥ 100 kg on Day 0 in Cohort 1 or brexucabtagene autoleucel at a targeted dose of 0.5 x 10^6 anti-CD19 CAR T cells/kg, with a maximum dose of 0.5 x 10^8 anti-CD19 CAR T cells for participants ≥ 100 kg on Day 0 in Cohort 2.
  Interventions: Biological: brexucabtagene autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Axicabtagene Ciloleucel

INTERVENTIONS:
Biological: brexucabtagene autoleucel — A single infusion of brexucabtagene autoleucel (KTE-X19) anti-CD 19 CAR T cells
  Other Names: KTE-X19, TECARTUS™
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously
Drug: Axicabtagene Ciloleucel — A single infusion of axicabtagene ciloleucel anti-CD 19 CAR T cells

SUMMARY:
The goal of this clinical study is to test how well the study drug, brexucabtagene autoleucel (KTE-X19), works in participants with relapsed/refractory (r/r) mantle cell lymphoma (MCL).

DETAILED DESCRIPTION:
Study KTE-C19-102 enrolled participants with r/r MCL who have been treated with up to 5 prior regimens including a Bruton's tyrosine kinase inhibitor (BTKi) in Cohort 1 and Cohort 2. However, to fulfill FDA Postmarketing Requirement, Cohort 3 is added to the study. It will include participants with r/r MCL who have been treated with up to 5 prior regimens but have not received prior therapy with a BTKi.

The primary analysis in Cohort 1 and Cohort 2 is already completed. Data for Cohort 3 will be analyzed separately. Therefore, details for Cohort 3 were registered separately (NCT04880434) on ClinicalTrials.gov as this cohort will not be part of the main study analysis.

After the end of KTE-C19-102, subjects who received an infusion of anti-CD19 CAR T cells will complete the remainder of the 15-year follow-up assessments in a separate long-term follow-up study, KT-US-982-5968

ELIGIBILITY:
Key Inclusion Criteria:

Up to 5 prior regimens for Mantle cell lymphoma. Prior therapy must have included:

* Anthracycline or bendamustine-containing chemotherapy and
* Anti-CD20 monoclonal antibody therapy and
* Ibrutinib or acalabrutinib

At least 1 measurable lesion

Platelet count ≥ 75,000/uL

Creatinine clearance (as estimated by Cockcroft Gault) > or = to 60 mL/min

Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings

Baseline oxygen saturation >92% on room air.

Key Exclusion Criteria:

* Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (HBsAG positive) or hepatitis C virus (anti-HCV positive). A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per standard serological and genetic testing
* History of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, cerebral edema, posterior reversible encephalopathy syndrome, or any autoimmune disease with central nervous system (CNS) involvement
* Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (32):
- United States (24):
  - Banner MD Anderson, Gilbert, Arizona
  - City of Hope, Duarte, California
  - University California Los Angeles (UCLA), Santa Monica, California
  - Stanford University, Stanford, California
  - Sarah Cannon, Denver, Colorado
  - University of Miami, Miami, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Robert W. Franz Cancer Research Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- France (3):
  - Centre Hospitalier Universitaire (CHU), Bordeaux
  - Hospital Saint Louis, Paris
  - Hopital Haut-Leveque, Pessac
- Germany (2):
  - Universitätsklinik Dresden, Dresden
  - Universitaetsklinikum Wuerzburg, Würzburg
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michael Wang,1 Javier Munoz,2 Andre Goy,3 Frederick L. Locke,4 Caron A. Jacobson,5 Brian T. Hill,6 John M. Timmerman,7 Houston Holmes,8 Samantha Jaglowski,9 Ian W. Flinn,10 Peter A. McSweeney,11 David B. Miklos,12 John M. Pagel,13 Marie José Kersten,14 Noel Milpied,15 Henry Fung,16 Max S. Topp,17 Roch Houot,18 Amer Beitinjaneh,19 Weimin Peng,20 Lianqing Zheng,20 John M. Rossi,20 Rajul K. Jain,20 Arati V. Rao,20 and Patrick M. Reagan21
- [Background] Wang M, Munoz J, Goy A, Locke FL, Jacobson CA, Hill BT, Timmerman JM, Holmes H, Jaglowski S, Flinn IW, McSweeney PA,Miklos DB, Pagel JM, Kersten MJ, Peng W,Zheng L,Rossi JM, Jain RK, Rao AV, Reagan PM
- [Background] Wang, Michael L., MD(1); Munoz, Javier, MD(2); Goy, Andre, MD(3); Locke, Frederick L., MD(4); Jacobson, Caron A., MD, MMSc(5); Hill, Brian T., MD(6); Timmerman, John M., MD(7); Holmes, Houston, MD(8); Jaglowski, Samantha, MD, MPH(9); Flinn, Ian W., MD, PhD(10); McSweeney, Peter A., MD(11); Miklos, David B., MD, PhD(12); Pagel, John M., MD, PhD, DSc(13); Jose Kersten, Marie, MD, PhD(14); Peng, Weimin, MS(15); Zheng, Lianqing, PhD(15); Rossi, John M., MS(15); Jain, Rajul K., MD(15); Rao, Arati V., MD(15); Reagan, Patrick M, MD(16)
- [Background] Wang, Michael; Lundry Locke, Frederick; Munoz, Javier; Goy, Andre; Eccleston Holmes, Houston; Siddiqi, Tanya; Flinn, Ian; McSweeney, Peter A; Michael Reagan, Patrick; Thomas Hill, Brian; Jacobson, Caron A.; Rizzieri, David A.; Heffner, Leonard T.; Mary Jaglowski, Samantha; Bernard Miklos, David; Shaughnessy, Paul; Unabia, Sherry; Rossi, John M.; Jiang, Yizhou; Jain, Rajul K.
- [Background] Cheah CY, Chihara D, Romaguera JE, Fowler NH, Seymour JF, Hagemeister FB, Champlin RE, Wang ML. Patients with mantle cell lymphoma failing ibrutinib are unlikely to respond to salvage chemotherapy and have poor outcomes. Ann Oncol. 2015 Jun;26(6):1175-1179. doi: 10.1093/annonc/mdv111. Epub 2015 Feb 23. PMID 25712454
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Dreyling M, Jurczak W, Jerkeman M, Silva RS, Rusconi C, Trneny M, Offner F, Caballero D, Joao C, Witzens-Harig M, Hess G, Bence-Bruckler I, Cho SG, Bothos J, Goldberg JD, Enny C, Traina S, Balasubramanian S, Bandyopadhyay N, Sun S, Vermeulen J, Rizo A, Rule S. Ibrutinib versus temsirolimus in patients with relapsed or refractory mantle-cell lymphoma: an international, randomised, open-label, phase 3 study. Lancet. 2016 Feb 20;387(10020):770-8. doi: 10.1016/S0140-6736(15)00667-4. Epub 2015 Dec 7. PMID 26673811
- [Background] Epperla N, Hamadani M, Cashen AF, Ahn KW, Oak E, Kanate AS, Calzada O, Cohen JB, Farmer L, Ghosh N, Tallarico M, Nabhan C, Costa LJ, Kenkre VP, Hari PN, Fenske TS. Predictive factors and outcomes for ibrutinib therapy in relapsed/refractory mantle cell lymphoma-a "real world" study. Hematol Oncol. 2017 Dec;35(4):528-535. doi: 10.1002/hon.2380. Epub 2017 Jan 8. PMID 28066928
- [Background] Fisher RI, Bernstein SH, Kahl BS, Djulbegovic B, Robertson MJ, de Vos S, Epner E, Krishnan A, Leonard JP, Lonial S, Stadtmauer EA, O'Connor OA, Shi H, Boral AL, Goy A. Multicenter phase II study of bortezomib in patients with relapsed or refractory mantle cell lymphoma. J Clin Oncol. 2006 Oct 20;24(30):4867-74. doi: 10.1200/JCO.2006.07.9665. Epub 2006 Sep 25. PMID 17001068
- [Background] Goy A, Sinha R, Williams ME, Kalayoglu Besisik S, Drach J, Ramchandren R, Zhang L, Cicero S, Fu T, Witzig TE. Single-agent lenalidomide in patients with mantle-cell lymphoma who relapsed or progressed after or were refractory to bortezomib: phase II MCL-001 (EMERGE) study. J Clin Oncol. 2013 Oct 10;31(29):3688-95. doi: 10.1200/JCO.2013.49.2835. Epub 2013 Sep 3. PMID 24002500
- [Background] Jain P, Kanagal-Shamanna R, Zhang S, Ahmed M, Ghorab A, Zhang L, Ok CY, Li S, Hagemeister F, Zeng D, Gong T, Chen W, Badillo M, Nomie K, Fayad L, Medeiros LJ, Neelapu S, Fowler N, Romaguera J, Champlin R, Wang L, Wang ML. Long-term outcomes and mutation profiling of patients with mantle cell lymphoma (MCL) who discontinued ibrutinib. Br J Haematol. 2018 Nov;183(4):578-587. doi: 10.1111/bjh.15567. Epub 2018 Sep 2. PMID 30175400
- [Background] Kratz A, Ferraro M, Sluss PM, Lewandrowski KB. Case records of the Massachusetts General Hospital. Weekly clinicopathological exercises. Laboratory reference values. N Engl J Med. 2004 Oct 7;351(15):1548-63. doi: 10.1056/NEJMcpc049016. No abstract available. PMID 15470219
- [Background] Lee DW, Gardner R, Porter DL, Louis CU, Ahmed N, Jensen M, Grupp SA, Mackall CL. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014 Jul 10;124(2):188-95. doi: 10.1182/blood-2014-05-552729. Epub 2014 May 29. PMID 24876563
- [Background] Locke FL, Ghobadi A, Jacobson CA, Miklos DB, Lekakis LJ, Oluwole OO, Lin Y, Braunschweig I, Hill BT, Timmerman JM, Deol A, Reagan PM, Stiff P, Flinn IW, Farooq U, Goy A, McSweeney PA, Munoz J, Siddiqi T, Chavez JC, Herrera AF, Bartlett NL, Wiezorek JS, Navale L, Xue A, Jiang Y, Bot A, Rossi JM, Kim JJ, Go WY, Neelapu SS. Long-term safety and activity of axicabtagene ciloleucel in refractory large B-cell lymphoma (ZUMA-1): a single-arm, multicentre, phase 1-2 trial. Lancet Oncol. 2019 Jan;20(1):31-42. doi: 10.1016/S1470-2045(18)30864-7. Epub 2018 Dec 2. PMID 30518502
- [Background] Martin P, Maddocks K, Leonard JP, Ruan J, Goy A, Wagner-Johnston N, Rule S, Advani R, Iberri D, Phillips T, Spurgeon S, Kozin E, Noto K, Chen Z, Jurczak W, Auer R, Chmielowska E, Stilgenbauer S, Bloehdorn J, Portell C, Williams ME, Dreyling M, Barr PM, Chen-Kiang S, DiLiberto M, Furman RR, Blum KA. Postibrutinib outcomes in patients with mantle cell lymphoma. Blood. 2016 Mar 24;127(12):1559-63. doi: 10.1182/blood-2015-10-673145. Epub 2016 Jan 13. PMID 26764355
- [Background] Rule S, Dreyling M, Goy A, Hess G, Auer R, Kahl B, Cavazos N, Liu B, Yang S, Clow F, Goldberg JD, Beaupre D, Vermeulen J, Wildgust M, Wang M. Outcomes in 370 patients with mantle cell lymphoma treated with ibrutinib: a pooled analysis from three open-label studies. Br J Haematol. 2017 Nov;179(3):430-438. doi: 10.1111/bjh.14870. Epub 2017 Aug 18. PMID 28832957
- [Background] Rule S, Dreyling M, Goy A, Hess G, Auer R, Kahl B, Hernandez-Rivas JA, Qi K, Deshpande S, Parisi L, Wang M. Ibrutinib for the treatment of relapsed/refractory mantle cell lymphoma: extended 3.5-year follow up from a pooled analysis. Haematologica. 2019 May;104(5):e211-e214. doi: 10.3324/haematol.2018.205229. Epub 2018 Nov 15. No abstract available. PMID 30442728
- [Background] Topp MS, Gokbuget N, Stein AS, Zugmaier G, O'Brien S, Bargou RC, Dombret H, Fielding AK, Heffner L, Larson RA, Neumann S, Foa R, Litzow M, Ribera JM, Rambaldi A, Schiller G, Bruggemann M, Horst HA, Holland C, Jia C, Maniar T, Huber B, Nagorsen D, Forman SJ, Kantarjian HM. Safety and activity of blinatumomab for adult patients with relapsed or refractory B-precursor acute lymphoblastic leukaemia: a multicentre, single-arm, phase 2 study. Lancet Oncol. 2015 Jan;16(1):57-66. doi: 10.1016/S1470-2045(14)71170-2. Epub 2014 Dec 16. PMID 25524800
- [Background] Wang M, Schuster SJ, Phillips T, Lossos IS, Goy A, Rule S, Hamadani M, Ghosh N, Reeder CB, Barnett E, Bravo MC, Martin P. Observational study of lenalidomide in patients with mantle cell lymphoma who relapsed/progressed after or were refractory/intolerant to ibrutinib (MCL-004). J Hematol Oncol. 2017 Nov 2;10(1):171. doi: 10.1186/s13045-017-0537-5. PMID 29096668
- [Background] Wang ML, Rule S, Martin P, Goy A, Auer R, Kahl BS, Jurczak W, Advani RH, Romaguera JE, Williams ME, Barrientos JC, Chmielowska E, Radford J, Stilgenbauer S, Dreyling M, Jedrzejczak WW, Johnson P, Spurgeon SE, Li L, Zhang L, Newberry K, Ou Z, Cheng N, Fang B, McGreivy J, Clow F, Buggy JJ, Chang BY, Beaupre DM, Kunkel LA, Blum KA. Targeting BTK with ibrutinib in relapsed or refractory mantle-cell lymphoma. N Engl J Med. 2013 Aug 8;369(6):507-16. doi: 10.1056/NEJMoa1306220. Epub 2013 Jun 19. PMID 23782157
- [Derived] Wang M, Munoz J, Goy A, Locke FL, Jacobson CA, Hill BT, Timmerman JM, Holmes H, Jaglowski S, Flinn IW, McSweeney PA, Miklos DB, Pagel JM, Kersten MJ, Bouabdallah K, Khanal R, Topp MS, Houot R, Beitinjaneh A, Peng W, Fang X, Shen RR, Siddiqi R, Kloos I, Reagan PM. Three-Year Follow-Up of KTE-X19 in Patients With Relapsed/Refractory Mantle Cell Lymphoma, Including High-Risk Subgroups, in the ZUMA-2 Study. J Clin Oncol. 2023 Jan 20;41(3):555-567. doi: 10.1200/JCO.21.02370. Epub 2022 Jun 4. PMID 35658525
- [Derived] Wang M, Jain P, Chi TL, Chen SE, Heimberger A, Weathers SP, Zheng L, Rao AV, Rossi JM. Management of a patient with mantle cell lymphoma who developed severe neurotoxicity after chimeric antigen receptor T-cell therapy in ZUMA-2. J Immunother Cancer. 2020 Oct;8(2):e001114. doi: 10.1136/jitc-2020-001114. PMID 33067318
- [Derived] Wang M, Munoz J, Goy A, Locke FL, Jacobson CA, Hill BT, Timmerman JM, Holmes H, Jaglowski S, Flinn IW, McSweeney PA, Miklos DB, Pagel JM, Kersten MJ, Milpied N, Fung H, Topp MS, Houot R, Beitinjaneh A, Peng W, Zheng L, Rossi JM, Jain RK, Rao AV, Reagan PM. KTE-X19 CAR T-Cell Therapy in Relapsed or Refractory Mantle-Cell Lymphoma. N Engl J Med. 2020 Apr 2;382(14):1331-1342. doi: 10.1056/NEJMoa1914347. PMID 32242358
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=KTE-C19-102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States, France, Netherlands and Germany.
Pre-assignment Details: Participants from 2 x 10^6 axicabtagene ciloleucel (AC) didn't contribute to primary and secondary analysis. The process used to manufacture axicabtagene ciloleucel was modified to manufacture brexucabtagene autoleucel (KTE-X19).
Groups:
- 2 x 10^6 Axicabtagene Ciloleucel: Participants with relapsed/refractory mantle cell lymphoma (MCL) received conditioning chemotherapy (CTE) consisting of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day intravenous (IV) infusion for 3 days followed by a single infusion of axicabtagene ciloleucel at a targeted dose of 2 x 10^6 anti-CD19 chimeric antigen receptor (CAR) T cells/kg on Day 0.
- Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel: Participants with relapsed/refractory MCL received CTE consisting of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day IV infusion for 3 days followed by a single infusion of brexucabtagene autoleucel at a targeted dose of 2 x 10^6 anti-CD19 CAR T cells/kg, with a maximum dose of 2 x 10^8 anti-CD19 CAR T cells for participants ≥ 100 kg on Day 0.
- Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel: Participants with relapsed/refractory MCL received conditioning chemotherapy consisting of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day IV infusion for 3 days followed by a single infusion of brexucabtagene autoleucel at a targeted dose of 0.5 x 10^6 anti-CD19 CAR T cells/kg, with a maximum dose of 0.5 x 10^8 anti-CD19 CAR T cells for participants ≥ 100 kg on Day 0.
Period: Overall Study
Arm/Group | 2 x 10^6 Axicabtagene Ciloleucel | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Started | 14 | 74 | 17
Safety Analysis Set (Treated Participants) | 10 | 68 | 14
Completed | 8 | 23 (Rolled over to another Long Term Follow Up (LTFU) study.) | 5 (Rolled over to another LTFU study.)
Not Completed | 6 | 51 | 12
Not completed — Death | 2 | 41 | 6
Not completed — Enrolled but never treated | 0 | 6 | 3
Not completed — Enrolled, did not initiate AC | 4 | 0 | 0
Not completed — Full consent withdrawal | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants treated with any dose of anti-CD19 CAR T cells.
Groups:
- 2 x 10^6 Axicabtagene Ciloleucel: Participants with relapsed/refractory MCL received CTE consisting of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day IV infusion for 3 days followed by a single infusion of axicabtagene ciloleucel at a targeted dose of 2 x 10^6 anti-CD19 CAR T cells/kg on Day 0.
- Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel: Participants with relapsed/refractory MCL received conditioning chemotherapy consisting of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day IV infusion for 3 days followed by a single infusion of brexucabtagene autoleucel at a targeted dose of 2 x 10^6 anti-CD19 CAR T cells/kg, with a maximum dose of 2 x 10^8 anti-CD19 CAR T cells for participants ≥ 100 kg on Day 0.
- Total: Total of all reporting groups
Arm/Group | 2 x 10^6 Axicabtagene Ciloleucel | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel | Total
Number analyzed (Participants) | 10 | 68 | 14 | 92
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 4 | 29 | 11 | 44
  >= 65 years | 6 | 39 | 3 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 3 | 15
  Male | 9 | 57 | 11 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 11 | 2 | 13
  Not Hispanic or Latino | 9 | 55 | 12 | 76
  Unknown or Not Reported | 1 | 2 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 0 | 1 | 0 | 1
  Race: White | 10 | 62 | 13 | 85
  Race: Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 1
  Race: Others | 0 | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  Netherlands | 0 | 2 | 0 | 2
  United States | 10 | 62 | 14 | 86
  France | 0 | 3 | 0 | 3
  Germany | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR) Per the Lugano Classification According to Independent Radiology Review Committee (IRRC) in Cohort 1
Description: OR: complete metabolic response(CMR),complete radiological response(CRR),partial MR response(PMR),partial RR(PRR).CMR:score 1(no uptake above background)/2(uptake ≤ mediastinum)/3(uptake > mediastinum but ≤ liver)with/without a residual mass on positron emission tomography 5-point scale;no new lesions.CRR:target nodes/nodal masses regressed to ≤ 1.5 cm in longest transverse diameter of lesion(LDi);no extralymphatic sites of disease;absent non-measured lesion(NMLs);organ enlargement regress to normal;no new sites;bone marrow normal by morphology. PMR:score 4(uptake moderately > liver)/5(uptake markedly > liver, new lesions)with reduced uptake compared with baseline and residual mass;no new lesions;responding disease at interim/residual disease at end of treatment (EOT).PRR: ≥ 50% decrease in sum of the product of the diameters(SPD)of up to 6 target measurable nodes and extra-nodal sites;absent/normal, regressed, but no increase of NMLs;spleen regressed by > 50% in length beyond normal.
Time Frame: Up to 7.8 years
Population: mITT set included all participants enrolled and treated with anti-CD19 CAR T cells at any dose in Cohort 1. Percentages were rounded off.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68
percentage of participants | 91

2. Primary Outcome: Percentage of Participants With Objective Response (OR) Per the Lugano Classification According to Independent Radiology Review Committee (IRRC) in Cohort 2
Description: OR: CMR, CRR, PMR, PRR. CMR: score 1(no uptake above background) / 2(uptake ≤ mediastinum) / 3(uptake > mediastinum but ≤ liver) with/without a residual mass on positron emission tomography 5-point scale; no new lesions. CRR: target nodes/nodal masses regressed to ≤ 1.5 cm in LDi; no extralymphatic sites of disease;absent non-measured lesion NMLs; organ enlargement regress to normal; no new sites; bone marrow normal by morphology. PMR: score 4(uptake moderately > liver) /5 (uptake markedly > liver, new lesions) with reduced uptake compared with baseline and residual mass; no new lesions; responding disease at interim/residual disease at EOT. PRR: ≥ 50% decrease in SPD of up to 6 target measurable nodes and extra-nodal sites; absent/normal, regressed, but no increase of NMLs; spleen regressed by > 50% in length beyond normal. Percentages were rounded off.
Time Frame: Up to 7.8 years
Population: The Modified intent to Treat (mITT) analysis set included all enrolled participants treated with any dose of anti-CD19 CAR T cells in Cohort 2
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 14
percentage of participants | 93

3. Secondary Outcome: Duration of Response (DOR) in Cohort 1 as Per Investigator Response
Description: DOR: time from the first OR to progressive disease (PD)/death. It is determined using Kaplan-Meier (KM) estimates. PD: score 4 (uptake moderately > liver)/ 5 (uptake markedly >liver and/or new lesions) with an increase in intensity of uptake from baseline; new fluorodeoxyglucose (FDG)-avid foci consistent with lymphoma at interim/EOT assessment; new FDG-avid foci consistent with lymphoma rather than another etiology; new/recurrent FDG-avid foci in bone marrow; an individual node/lesion must be abnormal with: LDi > 1.5 cm, increase by ≥ 50% from cross-product of LDi and perpendicular diameter (PPD) nadir, increase in LDi or shortest axis perpendicular to the LDi from nadir, the splenic length must increase by > 50% of the extent of its prior increase beyond baseline. If no prior splenomegaly, the increase must be ≥ 2 cm from baseline; new/recurrent splenomegaly; new or clear progression of pre-existing NMLs; new lesion; new/recurrent bone marrow involvement.
Time Frame: Up to 7.8 years
Population: Participants from the mITT analysis Set with objective response and available data in Cohort 1 were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 60
months | 36.5 [17.7 to 48.9]

4. Secondary Outcome: Duration of Response (DOR) in Cohort 2 as Per Investigator Response
Description: DOR: time from the first OR to PD/death. It is determined using KM estimates. PD: score 4 (uptake moderately > liver)/5 (uptake markedly >liver and/or new lesions) with an increase in intensity of uptake from baseline; new FDG-avid foci consistent with lymphoma at interim/EOT assessment; new FDG-avid foci consistent with lymphoma rather than another etiology; new/recurrent FDG-avid foci in bone marrow; an individual node/lesion must be abnormal with: LDi > 1.5 cm, increase by ≥ 50% from cross-product of LDi and PPD nadir, increase in LDi or shortest axis perpendicular to the LDi from nadir, the splenic length must increase by > 50% of the extent of its prior increase beyond baseline. If no prior splenomegaly, the increase must be ≥ 2 cm from baseline; new/recurrent splenomegaly; new or clear progression of pre-existing NMLs; new lesion; new/recurrent bone marrow involvement.
Time Frame: Up to 7.8 years
Population: Participants from the mITT analysis Set with objective response in Cohort 2 were analyzed. Participants not meeting the criteria for DOR at the time of data analysis were censored at their last evaluable disease assessment date.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 12
months | 57.5 [4.7 to NA] — Data for upper limit of CI is not available due to low number of participants with events.

5. Secondary Outcome: Percentage of Participants With Best Objective Response (BOR) as Per Investigator Assessment Determined by International Working Group (IWG) 2007 Criteria in Cohort 1
Description: BOR consists of (Complete response [CR], Partial response [PR], stable disease [SD], progressive disease [PD] and unknown). CR: disappearance of all detectable clinical evidence; PR: 50% decrease in the sum of the product of diameters (SPD) of up to 6 largest dominant nodal masses and >= 50% decrease in SPD of spleen/liver nodules; PD: appearance of any new lesions or >= 50% increase in SPD of more than one node or >= 50% increase in longest diameter of a previously identified node or >50% increase from nadir in the SPD of any previous lesions; SD: failure to attain CR/PR or PD. Percentages were rounded off.
Time Frame: Up to 7.8 years
Population: Participants from the mITT Analysis Set in Cohort 1 were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68
percentage of participants
  CR | 67.6 [55.2 to 78.5]
  PR | 20.6 [11.7 to 32.1]
  Stable disease | 8.8 [3.3 to 18.2]
  Progressive disease | 2.9 [0.4 to 10.2]

6. Secondary Outcome: Percentage of Participants With Best Objective Response (BOR) as Per Investigator Assessment Determined by Lugano Classification in Cohort 2
Description: BOR consists of CR (CMR/CRR), PR (PMR/PRR), SD, PD and not done. CMR/CRR and PMR/PRR are defined in Outcome Measure (OM) 1. PD is defined in OM 3. SD/no metabolic response (NMR): a score 4 (uptake moderately greater than [>] liver) or 5 (uptake markedly >liver and/ or new lesions) with no significant change in FDG uptake compared to baseline (screening), at an interim time point or end of treatment; no new sites of disease should be observed. Not done: no assessment at the time of analysis. Percentages were rounded off. Only categories with data are reported.
Time Frame: Up to 7.8 years
Population: Participants from the mITT Analysis Set in Cohort 2 were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 14
percentage of participants
  CR | 64.3 [35.1 to 87.2]
  PR | 21.4 [4.7 to 50.8]
  Stable disease | 7.1 [0.2 to 33.9]
  Not done | 7.1 [0.2 to 33.9]

7. Secondary Outcome: Percentage of Participants With Objective Response (OR) as Per Investigator Assessment Determined by International Working Group (IWG) 2007 Criteria in Cohort 1
Description: OR: CR or PR. CR: disappearance of all detectable clinical evidence; typically FDG-avid lymphoma (a post-treatment residual mass of any size is permitted if it is PET negative); variably FDG-avid lymphomas/FDG avidity unknown (all lymph nodes and nodal masses must have regressed to normal size); spleen and/or liver should be normal size and not be palpable; bone marrow aspirate and biopsy must show no evidence of disease. PR: 50% decrease in the SPD of up to 6 largest dominant nodal masses and ≥ 50% decrease in SPD of spleen/liver nodules; no increase in size of nodes, liver, or spleen and no new sites of disease; splenic and hepatic nodules must regress by ≥ 50% in the SPD; if participant has persistent bone marrow involvement and otherwise meets criteria for CR, will then be considered a PR; typically FDG-avid lymphoma (the post-treatment PET scan should be positive in at least 1 previously involved site. Percentages were rounded off.
Time Frame: Up to 7.8 years
Population: Participants from the mITT Analysis Set in Cohort 1 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68
percentage of participants | 88

8. Secondary Outcome: Percentage of Participants With Objective Response (OR) as Per Investigator Assessment Determined by Lugano Classification in Cohort 2
Description: OR: CMR, CRR, PMR, PRR. CMR: score 1(no uptake above background) / 2(uptake ≤ mediastinum) / 3(uptake > mediastinum but ≤ liver) with/without a residual mass on positron emission tomography 5-point scale; no new lesions. CRR: target nodes/nodal masses regressed to ≤ 1.5 cm in LDi ;no extralymphatic sites of disease;absent NMLs; organ enlargement regress to normal; no new sites;bone marrow normal by morphology. PMR: score 4 (uptake moderately > liver) /5 (uptake markedly > liver, new lesions) with reduced uptake compared with baseline and residual mass; no new lesions; responding disease at interim/residual disease at EOT. PRR: ≥ 50% decrease in SPD of up to 6 target measurable nodes and extra-nodal sites;absent/normal, regressed, but no increase of NMLs; spleen regressed by > 50% in length beyond normal. Percentages were rounded off.
Time Frame: Up to 7.8 years
Population: Participants from the mITT Analysis Set in Cohort 2 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 14
percentage of participants | 86

9. Secondary Outcome: Progression Free Survival (PFS) in Cohort 1 as Per Investigator Response.
Description: PFS was defined as the time from the brexucabtagene autoleucel infusion date to the date of PD or death from any cause. PD: a score 4 (uptake moderately > liver) or 5 (uptake markedly >liver and/or new lesions) with an increase in intensity of uptake from baseline; new FDG-avid foci consistent with lymphoma at interim or end of treatment assessment; new FDG-avid foci consistent with lymphoma rather than another etiology (eg, infection, inflammation); new or recurrent FDG-avid foci in bone marrow. PFS was determined using the KM estimates.
Time Frame: Up to 7.8 years
Population: Participants from the mITT Analysis Set in Cohort 1 were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68
months | 25.3 [12.7 to 42.8]

10. Secondary Outcome: Progression Free Survival (PFS) in Cohort 2 as Per Investigator Response.
Description: as for outcome 9
Time Frame: Up to 7.8 years
Population: Participants from the mITT Analysis Set in Cohort 2 were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 14
months | 29.5 [3.3 to NA] — Data for upper limit of CI is not available as the participants were censored.

11. Secondary Outcome: Overall Survival in Cohort 1
Description: Overall survival was defined as the time from brexucabtagene autoleucel infusion to the date of death from any cause. Overall survival was determined using the KM estimates.
Time Frame: Up to 7.8 years
Population: Participants from the mITT Analysis Set in Cohort 1 were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68
months | 46.5 [24.9 to 58.7]

12. Secondary Outcome: Overall Survival in Cohort 2
Description: as for outcome 11
Time Frame: Up to 7.8 years
Population: Participants from the mITT Analysis Set in Cohort 2 were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 14
months | NA [9.4 to NA] — Median and upper limit of CI were not reached due to low number of participants with events.

13. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial participants. The event did not necessarily have a relationship with study treatment. AE included worsening of a pre-existing medical condition. Worsening indicated that the pre-existing medical condition had increased in severity, frequency, and/or duration or had an association with a worse outcome. A pre-existing condition that had not worsened during the study or involved an intervention such as elective cosmetic surgery or a medical procedure while on study, was not considered an AE. TEAE was defined as any AE with onset on or after the start of treatment.
Time Frame: Up to 5 years
Population: Participants from the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
percentage of participants | 100 | 100

14. Secondary Outcome: Percentage of Participants With Decrease in Post-brexucabtagene Autoleucel Infusion Hematology Toxicity Values by Worst Toxicity Grade
Time Frame: Up to 5 years
Population: Participants from the Safety Analysis set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
percentage of participants
  Grade 3 or higher decrease in hemoglobin | 55.9 | 57.1
  Grade 3 or higher decrease in neutrophils | 98.5 | 100
  Grade 3 or higher decrease in platelets | 61.8 | 78.6
  Grade 3 or higher decrease in leukocytes | 98.5 | 92.9
  Grade 3 or higher decrease in lymphocytes | 95.6 | 100

15. Secondary Outcome: Percentage of Participants With Increase in Post-brexucabtagene Autoleucel Infusion Hematology Toxicity Values by Worst Toxicity Grade
Time Frame: Up to 5 years
Population: Participants from Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
percentage of participants
  Grade 3 or higher increase in leukocytes | 1.5 | 0
  Grade 3 or higher increase in lymphocytes | 1.5 | 0

16. Secondary Outcome: Percentage of Participants With Decrease in Post-brexucabtagene Autoleucel Infusion Chemistry Toxicity Values by Worst Toxicity Grade
Time Frame: Up to 5 years
Population: Participants from the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
percentage of participants
  Grade 3 or higher decrease in Potassium | 10.3 | 7.1
  Grade 3 or higher decrease in Calcium | 17.6 | 35.7
  Grade 3 or higher decrease in Magnesium | 0 | 0
  Grade 3 or higher decrease in Sodium | 13.2 | 28.6
  Grade 3 or higher decrease in Albumin | 7.4 | 7.1
  Grade 3 or higher decrease in Glucose | 1.5 | 7.1
  Grade 3 or higher decrease in Phosphate | 30.9 | 28.6

17. Secondary Outcome: Percentage of Participants With Increase in Post-brexucabtagene Autoleucel Infusion Chemistry Toxicity Values by Worst Toxicity Grade
Time Frame: Up to 5 years
Population: Participants from the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
percentage of participants
  Grade 3 or higher increase in Potassium | 0 | 0
  Grade 3 or higher increase in Calcium | 0 | 0
  Grade 3 or higher increase in Magnesium | 2.9 | 7.1
  Grade 3 or higher increase in Sodium | 4.4 | 0
  Grade 3 or higher increase in Alanine aminotransferase | 14.7 | 14.3
  Grade 3 or higher increase in Aspartate aminotransferase | 14.7 | 14.3
  Grade 3 or higher increase in Bilirubin | 1.5 | 0
  Grade 3 or higher increase in Creatinine | 5.9 | 7.1
  Grade 3 or higher increase in Urate | 16.2 | 21.4
  Grade 3 or higher increase in Direct bilirubin | 2.9 | 14.3
  Grade 3 or higher increase in Glucose | 5.9 | 21.4
  Grade 3 or higher increase in Alkaline phosphatase | 0 | 0

18. Secondary Outcome: Percentage of Participants With Anti-CD19 CAR Antibodies
Time Frame: Baseline up to Month 3
Population: Participants from the Safety Analysis Set were analyzed
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
percentage of participants | 21 | 21

19. Secondary Outcome: Maximum Number of CAR T Cells Measured Post-infusion
Time Frame: Up to Month 24
Population: Participants from the Safety Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
cells/μL | 313.02 (586.17) | 96.69 (109.33)

20. Secondary Outcome: Peak Serum Levels of C-Reactive Protein (CRP) in Blood
Description: Peak was defined as the maximum post-baseline level of the cytokine.
Time Frame: Baseline up to Week 4
Population: Participants from the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
mg/L | 4 [1 to 17] | 4 [1 to 8]

21. Secondary Outcome: Peak Serum Levels of C-X-C Motif Chemokine 10 (CXCL10), Granzyme B, Interferon-Gamma (IFN-γ), Interleukin-1 Receptor Antagonist (IL-1RA), Interleukin (IL)-2, IL-6, IL-7, IL-8,IL-10, IL-15, and Tumor Necrosis Factor-Alpha (TNF-α) in Blood
Description: Peak was defined as the maximum post-baseline level of the cytokine.
Time Frame: Baseline up to Week 4
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
pg/mL
  CXCL10 | 2000.00 [256.60 to 2000.00] | 2000.00 [495.80 to 2000.00]
  Granzyme B | 40.60 [1.00 to 6024.40] | 24.60 [1.00 to 231.70]
  IFN-gamma | 410.25 [7.50 to 1876.00] | 442.75 [7.50 to 1876.00]
  IL-1 RA | 1782.65 [158.40 to 9000.00] | 1783.05 [639.20 to 5012.20]
  IL-2 | 5.85 [0.90 to 77.60] | 6.70 [0.90 to 21.50]
  IL-6 | 86.00 [1.60 to 976.00] | 50.70 [3.20 to 976.00]
  IL-7 | 32.20 [16.30 to 72.80] | 31.80 [13.50 to 81.30]
  IL-8 | 41.19 [9.60 to 750.00] | 53.20 [10.60 to 140.70]
  IL-10 | 16.55 [0.70 to 246.10] | 246.10 [3.40 to 349.30]
  IL-15 | 40.30 [13.70 to 188.70] | 35.60 [27.10 to 80.90]
  TNF alpha | 9.50 [2.00 to 116.57] | 10.85 [2.60 to 62.50]

22. Secondary Outcome: Peak Serum Levels of Ferritin, Interleukin-2 Receptor Alpha (IL-2Rα), Intercellular Adhesion Molecule-1 (ICAM-1), Perforin, Vascular Cell Adhesion Molecule-1 (VCAM-1) in Blood
Description: Peak was defined as the maximum post-baseline level of the cytokine.
Time Frame: Baseline up to Week 4
Population: Participants from the Safety Analysis Set were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 68 | 14
ng/mL
  Ferritin | 1302.41 [0.80 to 25000] | 1126.52 [557.97 to 6177.17]
  IL-2 R alpha | 18.72 [2.20 to 100.00] | 23.95 [6.23 to 90.34]
  ICAM-1 | 1252.07 [230.12 to 60593.2467] | 1033.85 [218.96 to 1678.80]
  Perforin | 18.71 [0.69 to 100.00] | 13.84 [5.86 to 36.47]
  VCAM-1 | 1843.57 [503.80 to 156061.4308] | 1829.69 [416.85 to 3239.41]

23. Secondary Outcome: Percentage of Participants With Change Over Time in European Quality of Life-5 Dimensions(EQ-5D) Mobility Scale Score
Description: The European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) is a participant-answered questionnaire scoring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. For each dimension the participant is asked for a three-level assessment of their health on the current day: "no problems" (1), "some problems" (2), "extreme problems" (3). EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.11 (worst health state) to 1.00 (perfect health state). Positive numbers indicate improvement from baseline. The percentage of participants with each level of problem are reported. Percentages were rounded off.
Time Frame: Baseline, Week 4, Month 3, and Month 6
Population: Participants from the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 62 | 12
percentage of participants
  Baseline: No problems walking | 85 | 83
  Baseline: Slight problems walking | 11 | 17
  Baseline: Moderate problems walking | 3 | 0
  Baseline: Severe problems walking | 0 | 0
  Baseline: Unable to walk | 0 | 0
  Week 4: No problems walking: number analyzed (Participants) | 51 | 11
  Week 4: No problems walking | 49 | 73
  Week 4: Slight problems walking: number analyzed (Participants) | 51 | 11
  Week 4: Slight problems walking | 33 | 9
  Week 4: Moderate problems walking: number analyzed (Participants) | 51 | 11
  Week 4: Moderate problems walking | 6 | 18
  Week 4: Severe problems walking: number analyzed (Participants) | 51 | 11
  Week 4: Severe problems walking | 8 | 0
  Week 4: Unable to walk: number analyzed (Participants) | 51 | 11
  Week 4: Unable to walk | 4 | 0
  Month 3: No problems walking: number analyzed (Participants) | 55 | 11
  Month 3: No problems walking | 69 | 91
  Month 3: Slight problems walking: number analyzed (Participants) | 55 | 11
  Month 3: Slight problems walking | 18 | 9
  Month 3: Moderate problems walking: number analyzed (Participants) | 55 | 11
  Month 3: Moderate problems walking | 7 | 0
  Month 3: Severe problems walking: number analyzed (Participants) | 55 | 11
  Month 3: Severe problems walking | 4 | 0
  Month 3: Unable to walk: number analyzed (Participants) | 55 | 11
  Month 3: Unable to walk | 2 | 0
  Month 6: No problems walking: number analyzed (Participants) | 44 | 10
  Month 6: No problems walking | 75 | 90
  Month 6: Slight problems walking: number analyzed (Participants) | 44 | 10
  Month 6: Slight problems walking | 14 | 10
  Month 6: Moderate problems walking: number analyzed (Participants) | 44 | 10
  Month 6: Moderate problems walking | 7 | 0
  Month 6: Severe problems walking: number analyzed (Participants) | 44 | 10
  Month 6: Severe problems walking | 5 | 0
  Month 6: Unable to walk: number analyzed (Participants) | 44 | 10
  Month 6: Unable to walk | 0 | 0

24. Secondary Outcome: Percentage of Participants With Change Over Time in European Quality of Life-5 Dimensions(EQ-5D) Self-Care Scale Score
Description: as for outcome 23
Time Frame: Baseline, Week 4, Month 3, and Month 6
Population: Participants from the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 62 | 12
percentage of participants
  Baseline: No problems washing or dressing, | 95 | 100
  Baseline: Slight problems washing or dressing | 3 | 0
  Baseline: Moderate problems washing or dressing | 2 | 0
  Baseline: Severe problems washing or dressing | 0 | 0
  Baseline: Unable to wash or dress | 0 | 0
  Week 4: No problems washing or dressing,: number analyzed (Participants) | 52 | 11
  Week 4: No problems washing or dressing, | 67 | 91
  Week 4: Slight problems washing or dressing: number analyzed (Participants) | 52 | 11
  Week 4: Slight problems washing or dressing | 17 | 9
  Week 4: Moderate problems washing or dressing: number analyzed (Participants) | 52 | 11
  Week 4: Moderate problems washing or dressing | 4 | 0
  Week 4: Severe problems washing or dressing: number analyzed (Participants) | 52 | 11
  Week 4: Severe problems washing or dressing | 8 | 0
  Week 4: Unable to wash or dress: number analyzed (Participants) | 52 | 11
  Week 4: Unable to wash or dress | 4 | 0
  Month 3: No problems washing or dressing,: number analyzed (Participants) | 55 | 11
  Month 3: No problems washing or dressing, | 84 | 100
  Month 3: Slight problems washing or dressing: number analyzed (Participants) | 55 | 11
  Month 3: Slight problems washing or dressing | 11 | 0
  Month 3: Moderate problems washing or dressing: number analyzed (Participants) | 55 | 11
  Month 3: Moderate problems washing or dressing | 4 | 0
  Month 3: Severe problems washing or dressing: number analyzed (Participants) | 55 | 11
  Month 3: Severe problems washing or dressing | 2 | 0
  Month 3: Unable to wash or dress: number analyzed (Participants) | 55 | 11
  Month 3: Unable to wash or dress | 0 | 0
  Month 6: No problems washing or dressing,: number analyzed (Participants) | 44 | 10
  Month 6: No problems washing or dressing, | 93 | 100
  Month 6: Slight problems washing or dressing: number analyzed (Participants) | 44 | 10
  Month 6: Slight problems washing or dressing | 2 | 0
  Month 6: Moderate problems washing or dressing: number analyzed (Participants) | 44 | 10
  Month 6: Moderate problems washing or dressing | 0 | 0
  Month 6: Severe problems washing or dressing: number analyzed (Participants) | 44 | 10
  Month 6: Severe problems washing or dressing | 5 | 0
  Month 6: Unable to wash or dress: number analyzed (Participants) | 44 | 10
  Month 6: Unable to wash or dress | 0 | 0

25. Secondary Outcome: Percentage of Participants With Change Over Time in European Quality of Life-5 Dimensions(EQ-5D) Usual Activity Scale Score
Description: as for outcome 23
Time Frame: Baseline, Week 4, Month 3, and Month 6
Population: Participants from the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 65 | 12
percentage of participants
  Baseline: No problems doing usual activities | 82 | 75
  Baseline: Slight problems doing usual activities | 14 | 17
  Baseline: Moderate problems doing usual activities | 5 | 8
  Baseline: Severe problems doing usual activities | 0 | 0
  Baseline: Unable to do usual activities | 0 | 0
  Week 4: No problems doing usual activities: number analyzed (Participants) | 51 | 11
  Week 4: No problems doing usual activities | 43 | 36
  Week 4: Slight problems doing usual activities: number analyzed (Participants) | 51 | 11
  Week 4: Slight problems doing usual activities | 24 | 55
  Week 4: Moderate problems doing usual activities: number analyzed (Participants) | 51 | 11
  Week 4: Moderate problems doing usual activities | 22 | 9
  Week 4: Severe problems doing usual activities: number analyzed (Participants) | 51 | 11
  Week 4: Severe problems doing usual activities | 6 | 0
  Week 4: Unable to do usual activities: number analyzed (Participants) | 51 | 11
  Week 4: Unable to do usual activities | 6 | 0
  Month 3: No problems doing usual activities: number analyzed (Participants) | 56 | 11
  Month 3: No problems doing usual activities | 70 | 64
  Month 3: Slight problems doing usual activities: number analyzed (Participants) | 56 | 11
  Month 3: Slight problems doing usual activities | 16 | 36
  Month 3: Moderate problems doing usual activities: number analyzed (Participants) | 56 | 11
  Month 3: Moderate problems doing usual activities | 7 | 0
  Month 3: Severe problems doing usual activities: number analyzed (Participants) | 56 | 11
  Month 3: Severe problems doing usual activities | 4 | 0
  Month 3: Unable to do usual activities: number analyzed (Participants) | 56 | 11
  Month 3: Unable to do usual activities | 4 | 0
  Month 6: No problems doing usual activities: number analyzed (Participants) | 45 | 10
  Month 6: No problems doing usual activities | 73 | 70
  Month 6: Slight problems doing usual activities: number analyzed (Participants) | 45 | 10
  Month 6: Slight problems doing usual activities | 16 | 30
  Month 6: Moderate problems doing usual activities: number analyzed (Participants) | 45 | 10
  Month 6: Moderate problems doing usual activities | 9 | 0
  Month 6: Severe problems doing usual activities: number analyzed (Participants) | 45 | 10
  Month 6: Severe problems doing usual activities | 0 | 0
  Month 6: Unable to do usual activities: number analyzed (Participants) | 45 | 10
  Month 6: Unable to do usual activities | 2 | 0

26. Secondary Outcome: Percentage of Participants With Change Over Time in European Quality of Life-5 Dimensions(EQ-5D) Pain / Discomfort Activity Scale Score
Description: as for outcome 23
Time Frame: Baseline, Week 4, Month 3, and Month 6
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 65 | 12
percentage of participants
  Baseline: No pain or discomfort | 66 | 75
  Baseline: Slight pain or discomfort | 22 | 8
  Baseline: Moderate pain or discomfort | 9 | 17
  Baseline: Severe pain or discomfort | 3 | 0
  Baseline: Extreme pain or discomfort | 0 | 0
  Week 4: No pain or discomfort: number analyzed (Participants) | 54 | 11
  Week 4: No pain or discomfort | 63 | 64
  Week 4: Slight pain or discomfort: number analyzed (Participants) | 54 | 11
  Week 4: Slight pain or discomfort | 19 | 18
  Week 4: Moderate pain or discomfort: number analyzed (Participants) | 54 | 11
  Week 4: Moderate pain or discomfort | 19 | 18
  Week 4: Severe pain or discomfort: number analyzed (Participants) | 54 | 11
  Week 4: Severe pain or discomfort | 0 | 0
  Week 4: Extreme pain or discomfort: number analyzed (Participants) | 54 | 11
  Week 4: Extreme pain or discomfort | 0 | 0
  Month 3: No pain or discomfort: number analyzed (Participants) | 56 | 11
  Month 3: No pain or discomfort | 61 | 64
  Month 3: Slight pain or discomfort: number analyzed (Participants) | 56 | 11
  Month 3: Slight pain or discomfort | 16 | 27
  Month 3: Moderate pain or discomfort: number analyzed (Participants) | 56 | 11
  Month 3: Moderate pain or discomfort | 18 | 9
  Month 3: Severe pain or discomfort: number analyzed (Participants) | 56 | 11
  Month 3: Severe pain or discomfort | 4 | 0
  Month 3: Extreme pain or discomfort: number analyzed (Participants) | 56 | 11
  Month 3: Extreme pain or discomfort | 2 | 0
  Month 6: No pain or discomfort: number analyzed (Participants) | 46 | 10
  Month 6: No pain or discomfort | 65 | 70
  Month 6: Slight pain or discomfort: number analyzed (Participants) | 46 | 10
  Month 6: Slight pain or discomfort | 24 | 10
  Month 6: Moderate pain or discomfort: number analyzed (Participants) | 46 | 10
  Month 6: Moderate pain or discomfort | 9 | 20
  Month 6: Severe pain or discomfort: number analyzed (Participants) | 46 | 10
  Month 6: Severe pain or discomfort | 2 | 0
  Month 6: Extreme pain or discomfort: number analyzed (Participants) | 46 | 10
  Month 6: Extreme pain or discomfort | 0 | 0

27. Secondary Outcome: Percentage of Participants With Change Over Time in European Quality of Life-5 Dimensions(EQ-5D) Anxiety / Depression Activity Scale Score
Description: as for outcome 23
Time Frame: Baseline, Week 4, Month 3, and Month 6
Population: Participants from the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 65 | 12
percentage of participants
  Baseline: Not anxious or depressed | 75 | 67
  Baseline: Slight anxious or depressed | 20 | 33
  Baseline: Moderate anxious or depressed | 5 | 0
  Baseline: Severe anxious or depressed | 0 | 0
  Baseline: Extreme anxious or depressed | 0 | 0
  Week 4: Not anxious or depressed: number analyzed (Participants) | 54 | 11
  Week 4: Not anxious or depressed | 67 | 73
  Week 4: Slight anxious or depressed: number analyzed (Participants) | 54 | 11
  Week 4: Slight anxious or depressed | 26 | 27
  Week 4: Moderate anxious or depressed: number analyzed (Participants) | 54 | 11
  Week 4: Moderate anxious or depressed | 6 | 0
  Week 4: Severe anxious or depressed: number analyzed (Participants) | 54 | 11
  Week 4: Severe anxious or depressed | 2 | 0
  Week 4: Extreme anxious or depressed: number analyzed (Participants) | 54 | 11
  Week 4: Extreme anxious or depressed | 0 | 0
  Month 3: Not anxious or depressed: number analyzed (Participants) | 56 | 11
  Month 3: Not anxious or depressed | 70 | 91
  Month 3: Slight anxious or depressed: number analyzed (Participants) | 56 | 11
  Month 3: Slight anxious or depressed | 21 | 9
  Month 3: Moderate anxious or depressed: number analyzed (Participants) | 56 | 11
  Month 3: Moderate anxious or depressed | 9 | 0
  Month 3: Severe anxious or depressed: number analyzed (Participants) | 56 | 11
  Month 3: Severe anxious or depressed | 0 | 0
  Month 3: Extreme anxious or depressed: number analyzed (Participants) | 56 | 11
  Month 3: Extreme anxious or depressed | 0 | 0
  Month 6: Not anxious or depressed: number analyzed (Participants) | 46 | 10
  Month 6: Not anxious or depressed | 63 | 90
  Month 6: Slight anxious or depressed: number analyzed (Participants) | 46 | 10
  Month 6: Slight anxious or depressed | 26 | 10
  Month 6: Moderate anxious or depressed: number analyzed (Participants) | 46 | 10
  Month 6: Moderate anxious or depressed | 11 | 0
  Month 6: Severe anxious or depressed: number analyzed (Participants) | 46 | 10
  Month 6: Severe anxious or depressed | 0 | 0
  Month 6: Extreme anxious or depressed: number analyzed (Participants) | 46 | 10
  Month 6: Extreme anxious or depressed | 0 | 0

28. Secondary Outcome: Change Over Time in EQ-5D Visual Analogue Scale (VAS) Score
Description: EQ-5D is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-consists of two components: a health state profile and an optional visual analogue scale (VAS). The EQ5D-VAS records the participant's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. EQ-5D-VAS: range 0 to 100. A higher score indicates better self-reported health status. A positive change indicates an improvement.
Time Frame: Baseline, Week 4, Month 3, and Month 6
Population: Participants from the Safety Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on the scale
Arm/Group | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^6 Brexucabtagene Autoleucel
Number analyzed (Participants) | 65 | 12
scores on the scale
  Baseline | 82.0 (15.4) | 82.8 (16.1)
  Week 4: number analyzed (Participants) | 52 | 11
  Week 4 | 74.5 (15.6) | 71.4 (19.4)
  Month 3: number analyzed (Participants) | 56 | 11
  Month 3 | 80.2 (15.5) | 86.4 (11.0)
  Month 6: number analyzed (Participants) | 46 | 10
  Month 6 | 84.3 (16.9) | 89.9 (8.0)

ADVERSE EVENTS:
Time Frame: Adverse Event: Up to 5 years; All cause mortality: Up to 7.8 years
Description: Full Analysis Set included all enrolled participants. Safety Analysis Set included all participants treated with any dose of study drug. The Safety-Retreatment Analysis Set included all participants with re-treatment of KTE-X19 from Safety Analysis Set. All cause mortality was based on Full Analysis Set. SAE and other AE were based on the Safety Analysis Set.
Groups:
- Cohort 2: 0.5 x 10^8 Brexucabtagene Autoleucel: Participants with relapsed/refractory MCL received conditioning chemotherapy consisting of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day IV infusion for 3 days followed by a single infusion of brexucabtagene autoleucel at a targeted dose of 0.5 x 10^6 anti-CD19 CAR T cells/kg, with a maximum dose of 0.5 x 10^8 anti-CD19 CAR T cells for participants ≥ 100 kg on Day 0.
- Retreatment Cohort 1; Retreatment Cohort 2: Participants with relapsed/refractory MCL received a retreatment with conditioning chemotherapy consisting of fludarabine 30 mg/m^2/day and cyclophosphamide 500 mg/m^2/day IV infusion for 3 days followed by a single infusion of brexucabtagene autoleucel at a targeted dose of 2 x 10^6 anti-CD19 CAR T cells/kg, with a maximum dose of 2 x 10^8 anti-CD19 CAR T cells for participants ≥ 100 kg at Month 3.
Arm/Group | 2 x 10^6 Axicabtagene Ciloleucel | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel | Cohort 2: 0.5 x 10^8 Brexucabtagene Autoleucel | Retreatment Cohort 1 | Retreatment Cohort 2
All-Cause Mortality (participants affected / at risk) | 9/14 | 42/74 | 9/17 | 5/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 8/10 | 49/68 | 9/14 | 3/5 | 0/1
Other Adverse Events (participants affected / at risk) | 10/10 | 68/68 | 14/14 | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 x 10^6 Axicabtagene Ciloleucel (N=10) | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel (N=68) | Cohort 2: 0.5 x 10^8 Brexucabtagene Autoleucel (N=14) | Retreatment Cohort 1 (N=5) | Retreatment Cohort 2 (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatic haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis necrotising (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 14 | 2 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Corynebacterium infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Parvovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 12 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Salmonella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 4 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 3 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 4 | 12 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Communication disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 5 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 5 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Distributive shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 2 | 11 | 3 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nocardiosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 x 10^6 Axicabtagene Ciloleucel (N=10) | Cohort 1: 2 x 10^6 Brexucabtagene Autoleucel (N=68) | Cohort 2: 0.5 x 10^8 Brexucabtagene Autoleucel (N=14) | Retreatment Cohort 1 (N=5) | Retreatment Cohort 2 (N=1)
Anaemia (Blood and lymphatic system disorders) | 10 | 46 | 7 | 4 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 5 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 11 | 4 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 5 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 25 | 5 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 15 | 3 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 4 | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 6 | 1 | 0 | 0
Cardiac flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiomyopathy acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 4 | 9 | 2 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 21 | 5 | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 2 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 5 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 4 | 2 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 6 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 20 | 4 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 18 | 5 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 4 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 6 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 22 | 7 | 2 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 8 | 2 | 0 | 0
Asthenia (General disorders) | 3 | 13 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 7 | 27 | 6 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 7 | 26 | 7 | 1 | 0
Gait disturbance (General disorders) | 1 | 5 | 0 | 0 | 0
Generalised oedema (General disorders) | 1 | 2 | 2 | 0 | 0
Malaise (General disorders) | 1 | 5 | 3 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 3 | 1 | 0 | 0
Oedema (General disorders) | 1 | 4 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 15 | 5 | 1 | 0
Pain (General disorders) | 0 | 4 | 1 | 0 | 0
Pyrexia (General disorders) | 9 | 60 | 12 | 5 | 0
Swelling face (General disorders) | 0 | 0 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 12 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 3 | 1 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 4 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 5 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 6 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 10 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 21 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 14 | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 8 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 6 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 9 | 2 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 3 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 5 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 3 | 7 | 3 | 1 | 0
Neutrophil count decreased (Investigations) | 8 | 37 | 6 | 4 | 0
Platelet count decreased (Investigations) | 10 | 35 | 5 | 3 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 1 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 5 | 3 | 2 | 0 | 0
Weight increased (Investigations) | 0 | 5 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 8 | 28 | 7 | 3 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 15 | 7 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 13 | 4 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 23 | 4 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 19 | 4 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 21 | 5 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 10 | 4 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 22 | 4 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 25 | 4 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 8 | 3 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 8 | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 9 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7 | 2 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Aphasia (Nervous system disorders) | 2 | 9 | 4 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1 | 2 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 5 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 9 | 4 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 2 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 1 | 0 | 0
Dysgraphia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Encephalopathy (Nervous system disorders) | 2 | 12 | 2 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 7 | 25 | 5 | 1 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 2 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 5 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 3 | 5 | 2 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 6 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 3 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 7 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Tremor (Nervous system disorders) | 3 | 24 | 7 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 5 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 11 | 3 | 0 | 0
Communication disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 5 | 13 | 6 | 1 | 0
Depression (Psychiatric disorders) | 0 | 3 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 12 | 5 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 2 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 5 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 2 | 2 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 8 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 26 | 5 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 14 | 6 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 23 | 7 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 12 | 5 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 6 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 9 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 5 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Loss of personal independence in daily activities (Social circumstances) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 4 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 2 | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 14 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 30 | 10 | 3 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 2 | 1 | 0 | 0
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 10 | 0 | 0 | 0 | 0
Skin Infection (BILATERAL HANDS, IMPETIGO) (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Congestion (General disorders) | 1 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Papilloedema (Eye disorders) | 2 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Blood fibrinogen decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Past-pointing (Investigations) | 1 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Slow speech (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
General Disorder (General disorders) | 0 | 0 | 0 | 0 | 1 — Data has been reported as "General Disorder" term in the Retreatment Cohort 2 group for confidentiality reasons as there was only 1 participant in the group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Study Protocol: Amendment 6 (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT02601313/Prot_000.pdf
  • Study Protocol: Study Protocol: Amendment 9 (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT02601313/Prot_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan- Interim Results (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT02601313/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan- Final Results (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT02601313/SAP_003.pdf